CLINICAL TRIAL: NCT07247929
Title: Comparison of Postoperative Pain and Swelling in Flap Versus Flapless Technique for Surgical Removal of Partially Impacted Mandibular Third Molars: A Randomized Controlled Trial
Brief Title: Postoperative Pain and Swelling After Flap vsFlapless Technique For Mandibular Third Molar Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Watim Medical & Dental College (Other)
Responsible Party: Principal Investigator, Huma Bajar, prinicpal investigator, Watim Medical & Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMC-OMFS-FLAPvsFLAPLESS-2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Pain (Visceral, Somatic, or Neuropathic)
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flap technqiue (Experimental): Surgical extraction with mucoperiosteal flap elevation, bone guttering, tooth sectioning, and suturing.
  Interventions: Procedure: flap technqiue for mandibular third molar extraction Arm A
- flapless technquie (Experimental): Surgical extraction without flap elevation, minimal gingival reflection, bone guttering, and no suturing.
  Interventions: Procedure: flapless technquie arm b

INTERVENTIONS:
Procedure: flap technqiue for mandibular third molar extraction Arm A — Surgical extraction performed using a mucoperiosteal flap. A Ward's or modified Ward's incision is placed with a No. 15 blade. The flap is elevated to expose bone, followed by bone guttering with a straight fissure bur under saline irrigation. Tooth sectioning is carried out and fragments are removed. The socket is irrigated with saline and the flap is repositioned and sutured with 3-0 black braided silk.
  Arms: flap technqiue
Procedure: flapless technquie arm b — Surgical extraction of partially impacted mandibular third molar without raising a mucoperiosteal flap. Only minimal gingival reflection is performed using a periosteal elevator. Bone guttering and tooth sectioning are carried out using a bur under saline irrigation. Tooth fragments are removed. The socket is irrigated with saline and 0.2% chlorhexidine. No sutures are placed, and the site is allowed to heal by secondary intention
  Arms: flapless technquie

SUMMARY:
This randomized controlled trial evaluates postoperative pain and facial swelling following surgical removal of partially impacted mandibular third molars using flap versus flapless techniques. The aim is to determine which method results in lower postoperative morbidity on the second postoperative day.

DETAILED DESCRIPTION:
Impacted mandibular third molars frequently require surgical extraction, often involving mucoperiosteal flap elevation and bone removal. These steps may contribute to postoperative complications such as pain, swelling, and trismus. Minimally invasive alternatives, including flapless extraction, aim to reduce surgical trauma.

This study compares postoperative pain and swelling after flap versus flapless techniques in patients with partially impacted mesioangular mandibular third molars. Pain will be assessed using a 10-point Visual Analogue Scale (VAS), and swelling will be measured using standardized anthropometric facial measurements. A total of 160 participants will be randomized into two equal groups. All procedures will be performed by a single surgeon to reduce bias.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years

  * Either gender
  * Partially impacted mesioangular mandibular third molar confirmed clinically and radiographically
  * Second episode of pericoronitis
  * Swelling present on the affected side
  * No bone recession or periodontal disease on radiograph

Exclusion Criteria:

* HIV or HBV infection

  * Diabetes or other metabolic disorders
  * Bleeding disorders including von Willebrand disease, thalassemia, hemophilia, thrombocytosis, or thrombocytopenia
  * Periapical infection or acute pericoronitis at time of surgery
  * Severe trismus
  * Immunocompromised status

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | 2nd postoperative day
  Pain will be assessed on the 2nd postoperative day using the Visual Analogue Scale (VAS) ranging from 0 = no pain to 10 = worst pain. Patients will be instructed to rate their pain by marking a score on the 10-point VAS.
facial swelling measurement | 2nd postoperative day
  Measurements will be recorded in millimeters as:
  A = Gonion-Tragus B = Gonion-Outer canthus C = Gonion-Ala D = Gonion-Angle of mouth E = Gonion-Pogonion
  Total swelling = A + B + C + D + E. This method is described in the Operational Definition section of your synopsis.

CONTACTS AND LOCATIONS:
Locations (1):
- Watim Medical College&Dental Hospital, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No